CLINICAL TRIAL: NCT05421676
Title: Fetal Endoscopic Tracheal Occlusion (FETO) Trial for Congenital Diaphragmatic Hernia
Brief Title: Fetal Endoscopic Tracheal Occlusion for CDH (CDH)
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1724279
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Congenital Diaphragmatic Hernia; Fetal endoscopic tracheal occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FETO with GOLDBAL2 (Experimental): A balloon will be placed in the airway of the fetus during the FETO procedure.
  Interventions: Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100)

INTERVENTIONS:
Device: FETO with Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) — This will take place between gestation of 27w0d - 29w6d. The balloon will be removed at approximately 34 weeks gestation.

SUMMARY:
This is a single site pilot trial to assess the feasibility and safety of treating severe CDH with Fetal Endoscopic Tracheal Occlusion with the Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) at UC Davis Medical Center. The study will enroll pregnant women that meet study criteria. Participants will have placement of FETO between gestational age at 27 weeks plus 0 days and 29 weeks 6 days. The timing for removal of FETO will ideally be between 34 weeks 0 days and 34 weeks and 6 days but ultimately decided by the Fetal Diagnosis and Treatment Center at UC Davis Medical Center.

This study requires that study participants live within 30 minutes of the UC Davis Medical Center in order to maintain weekly follow up appointments while the balloon is in place and up to delivery. Additionally, there are lifestyle considerations where participants would be unable to carry on normal daily activities including exercise and sexual intercourse, not be able to work the remainder of the pregnancy, as well as have a support person that is available to stay with such as a spouse, friend, partner, parent.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability (meets psychosocial criteria below) for the duration of the study
3. Pregnant women, age 18 years and older
4. Singleton pregnancy
5. No pathogenic variants on microarray or pathologic findings on karyotype
6. Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects
7. Fetal CDH (left or right) with severe pulmonary hypoplasia, defined as o/e LHR <25% with liver up
8. Gestational age at FETO procedure: if o/e LHR <25% will be done at 27 weeks plus 0 days to 29 weeks plus 6 days
9. Meets psychosocial criteria

   * Willing to reside within 30 minutes of UC Davis Medical Center and ability to maintain follow up appointments
   * Patient has a support person (e.g. spouse, partner, friend, parent) that is available to stay with her for the duration of the pregnancy near the UC Davis Medical Center.
   * Willing to comply with restrictions of daily living including inability to exercise, have intercourse, or return to work

Exclusion Criteria:

1. Adults unable to consent
2. Prisoners
3. Multi-fetal pregnancy
4. History of latex allergy
5. History of preterm labor or incompetent cervix (requiring cerclage), short cervix (<20mm), or uterine anomaly predisposing to preterm labor
6. Psychosocial ineligibility

   * Inability to reside within 30 minutes of UC Davis Medical Center or inability to maintain follow up appointments
   * Social work will meet with each patient to evaluate the social situation and support system. Identifiable issues of social instability or compliance with the protocol will exclude her as a potential candidate.
7. Bilateral CDH, unilateral CDH with o/e LHR > 25% or unilateral CDH with o/e LHR <25% but liver completely down in abdomen
8. Additional fetal or genetic abnormalities that would impact care after delivery or be known to have an impact on outcome
9. Maternal contraindications to elective fetoscopic surgery
10. Significant placental abnormalities (abruption, chorioangioma, accreta) known at time of enrollment and/or surgery
11. Maternal isoimmunization or neonatal alloimmune thrombocytopenia
12. Maternal HIV, Hepatitis B with positive surface antigen, Hepatitis C with presence of virus in maternal blood due to risk of fetal transmission during the procedure
13. No safe or feasible fetoscopic approach to balloon placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of successful placements of the Goldballoon Detachable Balloon (GOLDBAL2) at gestational age 27 weeks zero days (27w0d) to 29 weeks and 6 days (29w6d) gestation. | 27 weeks 0 days to 29 weeks 6 days
  Success will be defined as completion with direct visual placement above the carina and confirmation on ultrasound done during the procedure.
Number of successful retrievals of the GOLDBAL2 | Removal prior to delivery approximately 34 weeks of gestation
  This will ideally occur around the 34th week of gestation and have the balloon removed prior to delivery.

SECONDARY OUTCOMES:
Change in observed to expected total fetal lung to head ratios (o/e TFLV) on prenatal magnetic resonance imaging (MRI) | baseline (prior to balloon placement), approximately 2 weeks after balloon retrieval
  Fetal MRI done prior to balloon placement and again done at approximately 2 weeks of balloon retrieval.
Change in fetal lung growth | baseline (before balloon placement), immediately prior to balloon retrieval
  Fetal ultrasounds will be done weekly while the balloon is in place. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR immediately prior to balloon removal.
Gestational age at delivery | At the time of delivery (up to approximately 34 weeks)
Survival of infant to hospital discharge or 180 days after hospitalized | Discharge from hospital or up to 180 days in the hospital
  This will be measured after the infant is delivered to hospital discharge or analyzed for survival at 180 days for those still hospitalized at that time point.
Number of maternal complications | up to 4-6 weeks postpartum
  Complications during pregnancy, and/or at delivery and follow-up to include; preterm labor, premature rupture of membranes (PROM), Preterm Premature Rupture of Membranes (PPROM), oligohydramnios, polyhydramnios, placental abruption, chorioamniotic separation, chorioamnionitis, and other infection.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT05421676/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT05421676/ICF_001.pdf